CLINICAL TRIAL: NCT02303938
Title: A Pilot Randomized Controlled Trial on the Feasibility and Efficacy of an Exercise Intervention to Improve Cognitive Functioning in Patients With Glioma
Brief Title: Effects of Exercise on Cognitive Function in Glioma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Responsible Party: Principal Investigator, Karin Gehring, Phd, Tilburg University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NL44024.008.13
Record Dates: First submitted 2013-07-15; First posted 2014-12-01 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Low Grade Glioma of Brain; Anaplastic Glioma of Brain
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- physical exercise (Experimental): Patients will exercise three times per week for 6 months home-based exercise intervention. Session duration will vary between 20 minutes and 45 minutes.
  Interventions: Behavioral: physical exercise
- Active control group (No Intervention): Patients in the active control group will be advised to walk regularly based on brochures from 30minutenbewegen.nl

INTERVENTIONS:
Behavioral: physical exercise — Patients in the intervention group will undergo a 6-month home-based exercise intervention. Patients will exercise (e.g., running, biking, swimming) three times per week for 6 months. Session duration will vary between 20 minutes and 45 minutes.
  Arms: physical exercise

SUMMARY:
The objective of this pilot randomized controlled trial (RCT) is to assess the feasibility and to determine the effect size of an exercise program in improving objective cognitive functioning.

DETAILED DESCRIPTION:
Clinical stable patients with 1) low grade glioma (LGG) or 2) anaplastic glioma under age 70 will undergo a home-based exercise program (intervention) or will be assigned to the active controle group. Patients in the intervention group will undergo a 6-month home-based exercise intervention. An individual exercise prescription will be based on the patients' level of aerobic fitness (VO2peak) as measured with cardiopulmonary testing (CPET; on a cycle ergometer with ECG and gas exchange measurement) at baseline. Patients will exercise (e.g., running, biking, swimming) three times per week for 6 months. Session duration will vary between 20 minutes and 45 minutes. Patients in the active control group will be advised to walk regularly based on brochures from 30minutenbewegen.nl.

All primary and secondary outcomes will be assessed at baseline (T0; prior to randomization), and at completion of the 6-month exercise intervention (T1), and at a similar time-point for patients in the active control group. These will include indicators of feasibility (accrual, adherence, compliance and attrition), subjective and objective physical fitness measures, neuropsychological performance scores, and self-reported cognitive symptoms and mental wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Grade II and III gliomas
* age < 50 years
* Karnofsky score > or equal 80
* clinically stable for a minimum of 6 months prior to study entry
* no recent anti-tumor treatment
* interested in undergoing a physical exercise program
* mild to moderate neuropsychological impairment based on normative comparison of objective test performance
* relative VO2peak that leaves room for further improvement of cardiorespiratory fitness.

Exclusion Criteria:

* patients with serious orthopedic conditions or motor deficits
* patients with serious cardiovascular, cardiopulmonary and neurological conditions (or risks)
* patients judged to have psychiatric (including alcohol and drug abuse)
* patients with severe cognitive problems
* patients who report to engage in vigorous exercise (≥7 METs) for more than 20 minutes on at least 3 days per week on a regular basis will be excluded

For assessment purposes, study participants will need to have basic fluency in the Dutch language.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
cognitive function as measured by neuropsychological tests | 6 months after the initial assessment
  neuropsychological test battery will be administered to patients at baseline and immediately after the intervention at 6 months

SECONDARY OUTCOMES:
Objective measures of physical fitness measured by cardiopulmonary exercise test (CPET) | 6 months after the initial assessment
  Intervention-related improvement of physical fitness will be assessed with a maximum cardiopulmonary exercise test (CPET). VO2 and of course adverse events are recorded immediately after the intervention ended at 6 months

OTHER OUTCOMES:
Patient reported outcome measured with self-reported questionnaires | 6 months after the initial assessment
  mood, sleep, fatique, quality of life, and depression are measured with self-reported questionaires at baseline and after intervention at 6 months such as Profile of Mood States (POMS) brief, Multidimensional Fatigue Inventory (MFI), Pittsburgh Sleep Inventory, MOS SF-36 Item Health Survey SF-36, and Brain-cancer specific HRQL questionnaire (QLQ-BN20)
Subjective cognition measured with Cognitive Functioning Scale (CFS) and Cognitive Failures Questionnaire (CFQ) | 6 months after the initial assessment
  Subjective cognition is measured with self-reported questionaire at baseline and after intervention at 6 months
Mental well-being measured with self-reported questionnaires | 6 months after the initial assessment
  Mental well-being is measured with specific questionaire at baseline and after intervention at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Karin Gehring, PhD, Principal Investigator — Tilburg University
Locations (1):
- Tilburg University, Tilburg, Nood-Brabant, Netherlands